CLINICAL TRIAL: NCT05008952
Title: Postprandial Triglycerides, Endothelial Function, and Inflammatory Cytokines as Potential Candidates for Early Risk Detection in Normal-weight Obesity
Brief Title: Identification of Early Cardiovascular Disease Risk Factors in Normal-weight Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: IRB-20-339-STW
Record Dates: First submitted 2021-08-04; First posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Metabolic Syndrome; Obesity
MeSH Terms: conditions — Metabolic Syndrome; Obesity

STUDY DESIGN:
Intervention Model Description: 3 study groups: control (normal body mass index, low body fat percentage), normal-weight obesity ((normal body mass index, high body fat percentage), and metabolic syndrome
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): The control group for this study will consist of individuals with normal BMI (18.5 - 24.9 kg/m2), body fat percent < 25% (male) or < 35% (female), and up to 1 other risk factor among the following: blood pressure > 130/85 mmHg, fasting glucose >100 mg/dL, fasting triglycerides >150 mg/dL, and HDL < 40 (male) or < 50 (female).
  Interventions: Other: High-fat shake
- Normal-weight obesity (Experimental): Individuals with normal-weight obesity will be defined as having normal BMI (18.5 - 24.9 kg/m2), body fat percent > 25% (male) or > 35% (female).
  Interventions: Other: High-fat shake
- Metabolic Syndrome (Active Comparator): Metabolic syndrome will be defined using the international Diabetes Federation criteria of an obese BMI ( > 30 kg/m2) and 2 or more of the following risk factors: blood pressure > 130/85 mmHg, fasting glucose >100 mg/dL, fasting triglycerides >150 mg/dL, and HDL < 40 (male) or < 50 (female).
  Interventions: Other: High-fat shake

INTERVENTIONS:
Other: High-fat shake — All participants will be given a high-fat test meal to examine their postprandial triglyceride response.

SUMMARY:
The purpose of this study is to identify early cardiovascular disease risk factors in those with "normal-weight obesity" (i.e., normal body, but high body fat percentage) that better track with their long-term cardiovascular disease risk.

ELIGIBILITY:
Inclusion Criteria:

Control group: normal BMI, body fat percentage < 25% for men and 35% for women

Normal-weight obesity group: normal BMI, body fat percentage > 25% for men and 35% for women

Metabolic syndrome group: BMI > 30 and 2 or more of the following: blood pressure >130/85 mmHg, fasting glucose >100 mg/dL, fasting triglycerides >150 mg/dL, HDL cholesterol < 40 mg/dL (men) or < 50 mg/dL (women).

Exclusion Criteria:

* Presence of pacemaker
* Pregnant
* use of tobacco products
* using lipid lowering drugs

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
4-hour triglycerides after fat tolerance test | Within 2 weeks of study enrollment
  Participants will undergo an abbreviated fat tolerance test, where fasting triglycerides are measured, a high-fat shake is consumed, and triglycerides measured once more 4 hours later. 4 hour triglycerides after the high-fat meal is our primary outcome.

SECONDARY OUTCOMES:
Flow-mediated dilation | Within 2 weeks of study enrollment
  Flow-mediated dilation is a non-invasive technique to investigate vascular health. This technique will be performed when participants are fasting and ~4 hours after the shake is completed (just before final measurement of triglycerides)
Fasting serum cytokines | Within 10 months of study enrollment
  A number of cytokines including GM-CSF, IFN-gamma, IL-1beta, IL-2, IL-5, IL-6, IL-8, IL-12p70, IL-13, IL-17, TNF-alpha, IL-4, IL-10 will be measured as additional cardiovascular disease risk factors.

CONTACTS AND LOCATIONS:
Locations (1):
- Oklahoma State University, Stillwater, Oklahoma, United States

REFERENCES:
- [Derived] Hart SM, Keirns BH, Sciarrillo CM, Malin SK, Kurti SP, Emerson SR. Cardiorespiratory fitness and submaximal exercise dynamics in normal-weight obesity and metabolically healthy obesity. Eur J Appl Physiol. 2024 Apr;124(4):1131-1142. doi: 10.1007/s00421-023-05344-8. Epub 2023 Nov 2. PMID 37917417